CLINICAL TRIAL: NCT05569850
Title: In Vivo Evaluation of Antibacterial Toothpaste Efficiency and Patients' Satisfaction: a Double-blind Randomised Controlled Trial
Brief Title: Efficacy of an Antibacterial Toothpaste and Patients' Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Collaborators: Unilever R&D (Industry)
Responsible Party: Principal Investigator, Lorenzo Breschi, Professor, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2.2022.
Record Dates: First submitted 2022-09-27; First posted 2022-10-06 (Actual); Results first posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Caries; Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Toothbrushing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recently introduced toothpaste (Experimental): Brushing twice a day with a recently introduced toothpaste.
  Interventions: Other: Brushing
- Commercial toothpaste (Active Comparator): Brushing twice a day with a commercially available toothpaste.
  Interventions: Other: Brushing

INTERVENTIONS:
Other: Brushing — Brushing the teeth 2x a day for 4 weeks.

SUMMARY:
The primary objective of this randomized controlled clinical trial (RCCT) will be to compare the efficacy in reducing the quantity of Streptococcus mutans (S. Mutans) in saliva of a recently introduced toothpaste compared to a commercially available toothpaste. The secondary outcomes will be to assess patients' impression of the toothpastes (in terms of taste, satisfaction etc.), and to investigate potential changes in dentin hypersensitivity, plaque formation and gingival inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with minimum 20 teeth;
2. Good oral hygiene level (gingival bleeding index not exceeding 20%)
3. Patients willing to participate in the study and able to sign an informed consent

Exclusion Criteria:

1. Tooth anomalies (amelogenesis imperfecta, dentinogenesis imperfecta etc.);
2. Intrinsic stain (fluorosis);
3. Caries lesions;
4. Advanced periodontal disease (probing >2, spontaneous gum bleeding, tooth mobility >1);
5. Smokers;
6. Use of orthodontic devices;
7. Use of antibiotics in the last 3 months;
8. Use of antibacterial mouth rinses in the last 3 months;
9. Potential allergies;
10. Drug and alcohol abuse;

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- DIBINEM, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Recently Introduced Toothpaste | Commercial Toothpaste
Started | 50 | 50
Completed | 46 | 39
Not Completed | 4 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Recently Introduced Toothpaste | Commercial Toothpaste | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.7 (0.3) | 25.3 (0.4) | 25.5 (0.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 55
  Male | 21 | 24 | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Potential patients were recruited through local advertisement or on-site, during routine dental check-ups within the Dental Clinic (DIBINEM, University of Bologna, Italy). Population: There was a drop-out of patients.
  participants
    Italy: number analyzed (Participants) | 46 | 39 | 85
    Italy | 46 | 39 | 85

OUTCOME MEASURES:

1. Primary Outcome: Bacterial Count of Streptococcus Mutans (S. Mutans)
Description: Agar Mitis salivarius with tellurium and bacitracin (MSTB) will be used for S. mutans isolation. The 0.1 ml saliva sample will be diluted with 0.9 ml of sterile normal saline; next, decimal dilutions of saliva will be made up to 10-3. Each medium plate will be cultured from 0.1 ml of the previously diluted sample to 10-3; then, the sample will be uniformly spread on the agar plates. Finally, the plates will be sealed. They will be incubated for 48 hours at 37°C. The bacterial colonies will be observed under a stereo microscope and identified by morphology and color. The CFU will be multiplied by the number of times the sample was originally diluted and expressed as the number of colony forming units per millilitre (CFU/mL) of saliva.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: log CFU/ml
Arm/Group | Recently Introduced Toothpaste | Commercial Toothpaste
Number analyzed (Participants) | 46 | 39
log CFU/ml | 4.261 (0.0867) | 4.277 (0.0931)

2. Secondary Outcome: Plaque Index
Description: The plaque will be disclosed using a disclosing solution and recorded as follows: score 0 = absence of plaque; score 1 = separate flecks of plaque on the cervical margin; score 2 = a thin, continuous band of plaque [up to 1 mm] at the cervical margin of the tooth; score 3 = a band of plaque wider than 1 mm, but covering less than one-third of the tooth crown; score 4 = plaque covering at least one-third, but less than two-third of the crown of the tooth; score 5 = plaque covering 2/3-crown or more of the crown of the tooth.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Recently Introduced Toothpaste | Commercial Toothpaste
Number analyzed (Participants) | 46 | 39
score on a scale | 0.1 (0.05) | 0.17 (0.1)

3. Secondary Outcome: Gingival Index
Description: A North Carolina periodontal probe (Hu-Friedy, Chicago, IL, USA) will be used for determine gingival index according to the following scale: score 0 = absence of inflammation; score 1 = mild inflammation-slightly slight change in color and little change in texture; score 2 = moderate inflammation-moderate glazing, redness, edema, and hypertrophy; score 3 = severe inflammation-marked redness and hypertrophy.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Recently Introduced Toothpaste | Commercial Toothpaste
Number analyzed (Participants) | 46 | 39
score on a scale | 0 (0) | 0 (0)

4. Secondary Outcome: Dentin Hypersensitivity
Description: Patients with self-reported dentin hypersensitivity will be considered. A 1-s air blast from approximately 1 cm distance will be applied onto exposed dentine. The participant's response will be assessed using the 4-point Schiff Sensitivity Scale (from 0: participant does not respond, to 3: participant responds to stimulus, considers it painful, and requests discontinuation;
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Recently Introduced Toothpaste | Commercial Toothpaste
Number analyzed (Participants) | 46 | 39
units on a scale | 0.19 (0.1) | 0.2 (0.1)

5. Secondary Outcome: Tooth Colour
Description: Participants' satisfaction before and after treatment will be recorded and the difference will be assessed. In order to obtain the data concerning patients' satisfaction with tooth color, a questionnaire containing aesthetic numeric visual-analogue scale ranging from 1 to 10 will be given to the subjects.
  1 = "Not satisfied at all" and 10 = "Very satisfied"
Time Frame: 4 weeks
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Recently Introduced Toothpaste | Commercial Toothpaste
Number analyzed (Participants) | 46 | 39
units on a scale | 8 (0.5) | 7.8 (0.5)

ADVERSE EVENTS:
Time Frame: Up to 4 weeks.
Arm/Group | Recently Introduced Toothpaste | Commercial Toothpaste
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT05569850/Prot_SAP_000.pdf
  • Informed Consent Form (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT05569850/ICF_001.pdf